CLINICAL TRIAL: NCT06463925
Title: Evaluation of Effaclar Duo+M on Inflammatory and Non-Inflammatory Lesions in Subjects With Mild to Moderate Acne on Face and Trunk (Back and Chest)
Brief Title: Evaluation of Effaclar Duo+M on Acne Lesions in Subjects With Mild to Moderate Acne on Face and Trunk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LRP23014-2223CBCL059 Effaclar
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Acne
Keywords: facial and truncal acne; Effaclar Duo+M; acne lesions
MeSH Terms: conditions — Acne Vulgaris; Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acneic participants group (Other): subjects with mild to moderate facial and truncal acne
  Interventions: Other: acneic participants group

INTERVENTIONS:
Other: acneic participants group — Application of Effaclar Duo+M to the face and trunk twice daily (morning and evening) after washing with the cleansing gel.

SUMMARY:
This single-center, open, non-randomized study aims the efficacy evaluation of Effaclar Duo+M and Effaclar+M Purifying foaming gel on total acne lesion count, pigmented lesions and scars for 6 months in subjects with mild to moderate facial and truncal acne.

DETAILED DESCRIPTION:
The study will be conducted in accordance with the principles of Resolution 466/2012 of the Conselho Nacional de Saúde do Brasil3, ethical principles from the Declaration of Helsinki (and subsequent modifications) and Good Clinical Practice.

Statistical methodology:

Quantitative variables, or those that can reasonably be treated as such, are summarized using the minimum, maximum, measures of central tendency such as the mean and median & measures of dispersion such as the standard deviation (SD). Qualitative variables are summarized in the form of counts and percentages.

Significance level:

The null hypothesis will generally be rejected if a p-value less than 0.05 (5% significance level) is produced by the statistical procedure.

ELIGIBILITY:
Inclusion Criteria:

* phototype I to VI
* mild to moderate acne on the face and trunk

Exclusion Criteria:

* cutaneous pathology on the studied zone other than acne
* topical or systemic treatment during the previous weeks liable to interfere with the assessment of the acceptability and efficacy of the studied products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
efficacy on total acne lesion count on face and trunk | from baseline to Day168
  The counting is performed by region (back, chest, face, total) and type of lesion (post-inflammatory hyperpigmentation, post-inflammatory erythema, scars, pustules, nodules, papules, closed comedones, open comedones.

SECONDARY OUTCOMES:
Evaluation of the degree of severity of acne on the face | from baseline to Day168
  Evaluation performed thanks to the Global Evaluation Acne (GEA) scale on a 6-point score: from 0 (Clean. No lesions) to 5 (Very severe).
Evaluation of the degree of severity of acne on the trunk | from baseline to Day168
  Evaluation performed thanks to the Investigator Global Assessment (IGA) scale on a 6-point score: from 0 (Absent) to 5 (Very serious).

CONTACTS AND LOCATIONS:
Overall Officials: Renato Moura, Principal Investigator — Centre International de Développement Pharmaceutique (CIDP)
Locations (1):
- CIDP Brasil, Rio de Janeiro, Brazil